CLINICAL TRIAL: NCT05070715
Title: Comparison of Microplastic Levels in Placenta and Cord Blood Samples of Pregnant Women With Fetal Growth Retardation and Healthy Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: Kutahya HSU
Record Dates: First submitted 2021-10-06; First posted 2021-10-07 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-10

CONDITIONS: Microplastic Levels in Placenta and Cord Blood

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Placental tissue and cord blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: FGR group: Estimated fetal weight <10th percentile
  Interventions: Other: Analyzing of microplastic level
- Group 2: Control group: Healthy pregnants who will give birth 37th and after gestational week
  Interventions: Other: Analyzing of microplastic level

INTERVENTIONS:
Other: Analyzing of microplastic level — Blood samples will be taken from the vein of the umbilical cord. Placental tissues will be taken from the maternal side of the placenta. Placental tissues and serum samples will be stored in the temperature set to -80 °C until analysis. Extraction methods involving chemical reactions will be used to separate and purify microplastics in placenta and cord blood samples. After the extraction process, analysis of microplastic levels in tissues and serum will be done by µ-Raman spectroscopy.

SUMMARY:
In this study, microplastic levels in the placenta and cord blood of pregnant women with fetal growth retardation and healthy pregnant women will be compared in placenta and cord blood samples after delivery.

DETAILED DESCRIPTION:
The study will be conducted with a total of 40 pregnant women, 20 of whom are in the control groups and those with FGR diagnoses. Cases in both groups will be matched in terms of demographic information. Demographic information (including socioeconomic status, educational level, region of residence), ultrasound and Doppler examination results, newborn weight at birth, APGAR score, gender, mode of delivery, whether there is a need for neonatal intensive care or not will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-40 years
* Gestational age between 320/7 - 396/7 weeks
* Singleton pregnancy
* For the FGR group: estimated fetal weight <10th percentile
* For the control group: being healthy pregnant
* Intact amniotic membrane

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: * Multiple pregnancies
  * Cardiovascular disease
  * Chronic hypertension
  * Autoimmune disease
  * Intrahepatic cholestasis of pregnancy
  * Preeclampsia-eclampsia
  * Sepsis
  * Placenta accreta spectrum
  * Abnormalities of placenta
  * The chromosomal or congenital structural anomaly of the fetus
  * Smoking
  * BMI >30 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-29 (Estimated); Primary Completion 2023-02-26 (Estimated); Study Completion 2023-03-26 (Estimated)

PRIMARY OUTCOMES:
Analyzing of microplastic levels in the placenta and cord blood of pregnant women | 1 year
  Microplastic levels in pregnant women's placenta and cord blood will be measured in placenta and cord blood samples after delivery.

SECONDARY OUTCOMES:
Investigation of the effect of microplastic level in placenta and cord blood on FGR | 1 month
  If there is a significant difference in other data, including the microplastic level, in the FGR group, the effect of each factor on the development of FGR will be analyzed by multi logistic regression analysis. In addition, if the microplastic level is found to be significantly higher in the FGR group, the cut-off value will be obtained by ROC analysis.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ragusa A, Svelato A, Santacroce C, Catalano P, Notarstefano V, Carnevali O, Papa F, Rongioletti MCA, Baiocco F, Draghi S, D'Amore E, Rinaldo D, Matta M, Giorgini E. Plasticenta: First evidence of microplastics in human placenta. Environ Int. 2021 Jan;146:106274. doi: 10.1016/j.envint.2020.106274. Epub 2020 Dec 2. PMID 33395930
- [Result] Braun T, Ehrlich L, Henrich W, Koeppel S, Lomako I, Schwabl P, Liebmann B. Detection of Microplastic in Human Placenta and Meconium in a Clinical Setting. Pharmaceutics. 2021 Jun 22;13(7):921. doi: 10.3390/pharmaceutics13070921. PMID 34206212